CLINICAL TRIAL: NCT00629187
Title: Phase I Dose Escalation Study of Temozolomide With Autologous Stem Cell Rescue for Patients With Relapsed/Refractory CNS Malignancy Including Isolated Metastatic Disease
Brief Title: Safety Study of High Dose Temozolomide to Treat Relapsed/Refractory Central Nervous System (CNS) Malignancy
Acronym: CN-306
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to lack of adequate enrollment.
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN-306
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Central Nervous System Neoplasms; Neoplasm Metastasis
Keywords: Lung Neoplasm; Breast Neoplasm; Melanoma; Central Nervous System Neoplasms; Neoplasm Metastasis; Neoplasm Second Primary; Peripheral Blood Stem Cell Transplantation
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Lung Neoplasms; Breast Neoplasms; Melanoma; Neoplasms, Second Primary | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Before taking part in this study, subjects will have stem cells collected in a procedure called apheresis. Once on this study, subjects will be admitted to the hospital and receive daily doses of temozolomide by mouth for 5 days. Stem cells will be given back to subjects who will remain in the hospital until blood counts have recovered. Doses of temozolomide will range from 350 mg to 1500 mg/m(squared) daily for 5 days (total dose 1750 to 7500 mg/m(squared).
  Other Names: Temodar

SUMMARY:
The goal of this study is to find the maximum dose of a drug, temozolomide, that can safely be given to subjects with brain tumors. Past studies showed that the maximum dose of temozolomide was limited by low blood counts. The investigators will use blood stem cells collected from bone marrow to help subjects recover their blood counts, a procedure called autologous stem cell transplant or stem cell rescue. This way, the investigators expect to be able to safely deliver very high doses of temozolomide. This study is only available at Tufts Medical Center.

DETAILED DESCRIPTION:
High dose chemotherapy and autologous stem cell transplant is an accepted treatment alternative for patients with brain tumors. Temozolomide has been approved for use by the United States Food and Drug Administration (FDA) for certain tumors of the brain. The doses of temozolomide given in this study will be higher than approved by the FDA and higher than those given in any prior studies.

Over 25 subjects will be enrolled on this study over a period of 5 years. This study will only be available at Tufts Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients or their health care proxies must be able to provide consent to participate in this trial.
* Patients must have one of the following diagnoses which has not responded or recurred following at least one prior chemotherapy regimen or radiation therapy:

  * anaplastic astrocytoma, glioblastoma multiforme or oligodendroglioma
  * primary CNS lymphoma
  * malignant disease metastatic to the CNS
* Patients must be candidates for high dose chemotherapy and autologous stem cell transplant according to the following criteria:

  * Patients must be between the ages of 18 and 70 years (inclusive)
  * Patients must have a left ventricular ejection fraction greater than or equal to 45% by MUGA or echocardiogram
  * Patients must have adequate pulmonary function with FEV1, FVC and DLCO greater than or equal to 50% of predicted
  * Patients must have serum direct bilirubin less than or equal to 2.0 mg/dl and transaminases less than or equal to 3x institutional upper limit of normal
  * Patients must have serum creatinine less than or equal to 2 mg/dl with creatinine clearance greater than or equal to 60 ml/min (either calculated or measured)
  * Patients must have an ECOG performance status between 0 and 2
* Patients must be at least 4 weeks from last cytoreductive chemotherapy.
* Expected survival of at least 3 months

Exclusion Criteria:

* Patients with uncontrolled metastatic disease outside of the CNS which would itself, in the investigator's opinion, limit survival to less than 6 months
* Patients with uncontrolled seizures are ineligible.
* Patients with a history of myocardial infarction within the preceding 6 months, significant arrhythmia within the preceding 3 months, or uncontrolled hypertension or congestive heart failure are ineligible.
* Patients with unstable angina are ineligible.
* Pregnant or lactating women are ineligible.
* Male and female patients who do not agree to practice approved methods of birth control for the duration of the study are ineligible.
* Patients with uncontrolled, active infection are ineligible.
* Patients infected with HIV are ineligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of temozolomide with hematopoietic stem cell rescue in patients with recurrent CNS malignancy | 5 years

SECONDARY OUTCOMES:
Estimate the response rate, response duration and survival according to established response definitions | 5 years
Determine the pharmacokinetics of high daily dosing of temozolomide in the transplant setting | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Klein, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States